CLINICAL TRIAL: NCT04557228
Title: Targeting ADAM17 Activity for Correction of Vascular Insulin Resistance in Type 2 Diabetes
Brief Title: ADAM17 and Vascular Function in Diabetes
Acronym: ADAM17
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Luis Martinez-Lemus, DVM, PhD, Professor in Medical Pharmacology Physiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025921
Record Dates: First submitted 2020-09-08; First posted 2020-09-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: endothelial dysfunction; vascular function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Phosphatidylserines

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded design with 34 subjects
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Study participants will receive 4 weeks of supplementation with 900mg placebo supplements
  Interventions: Dietary Supplement: Placebo
- Phosphatidylserine Supplementation (Experimental): Study participants will receive 4 weeks of supplementation with 900mg phosphatidylserine supplements.
  Interventions: Dietary Supplement: Phosphatidylserine

INTERVENTIONS:
Dietary Supplement: Placebo — 4 weeks of placebo supplements
  Arms: Placebo
Dietary Supplement: Phosphatidylserine — 4 weeks of phosphatidylserine supplements
  Arms: Phosphatidylserine Supplementation

SUMMARY:
The objective of this project is to determine the extent to which administration of the dietary supplement phosphatidylserine (PS), a competitive inhibitor of ADAM17 sheddase activity, effects vascular function and insulin-stimulated leg blood flow in subjects with T2D.

DETAILED DESCRIPTION:
As part of a randomized (1:1, experimental/placebo), double-blinded parallel design, each of the 34 subjects will complete 4 weeks (+/-4 days) of supplementation with either 900mg of a PS supplement or placebo. Assessment visits (2) will occur pre-intervention and post-intervention and include: 24-hour ambulatory blood pressure measurement (ABPM), Vitals, DEXA scan for body composition, fasting blood work, carotid-femoral pulse wave velocity (cfPWV), brachial and femoral artery FMDs, Femoral blood flow imaging during passive leg movement (PLM), glycocalyx integrity assessment via Glycocheck, and an oral glucose tolerance test (OGTT) with blood flow measurements and beat-to-beat sphygmomanometry via Finometer.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with a BMI of 25-39 kg/m2, who are 45-64 years of age at randomization.
2. T2D patients classified based on physician diagnosis.
3. No vulnerable populations (e.g., prisoners, pregnant, children) will be enrolled.

Exclusion Criteria:

1. Cardiovascular disease including myocardial infraction, heart failure, coronary artery disease, stroke
2. History of chronic renal or hepatic disease
3. Active cancer
4. Autoimmune diseases
5. Immunosuppressant therapy
6. Hormone replacement therapy
7. Excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
8. Current tobacco use
9. Pregnancy
10. Bodyweight change ≥5% within the last 6 months

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin-stimulated blood flow | baseline and 4 weeks
  Measure of blood flow during oral glucose tolerance test. Leg blood flow measures will be performed non-invasively via Ultrasound.

SECONDARY OUTCOMES:
Change in Vascular function | Baseline and 4 weeks
  Flow mediated dilation (FMD) in arm and passive limb movement (PLM) in the leg. Blood flow measures will be performed non-invasively via Ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri- NextGen Clinical Translational Science Unit, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT04557228/ICF_000.pdf